CLINICAL TRIAL: NCT04277416
Title: Survivorship and Effectiveness of the Ortho Development® Entrada™ Hip System for Total Hip Arthroplasty: A Prospective Multi-Centre Cohort Study
Brief Title: Survivorship and Effectiveness of the Ortho Development® Entrada™ Hip System for Total Hip Arthroplasty
Status: Enrolling by invitation | Type: Observational
Sponsor: Ortho Development Corporation (Industry)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: P-19-0055
Record Dates: First submitted 2019-11-06; First posted 2020-02-20 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Total Hip Replacement; Total Hip Arthroplasty
Keywords: Ortho Development; Entrada Hip System
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Entrada Hip System: All orthopaedic patients that are scheduled to undergo primary total hip arthroplasty using the Entrada™ Hip System within 12 weeks will be screened for the following eligibility criteria.
  Interventions: Device: Total Hip Arthroplasty

INTERVENTIONS:
Device: Total Hip Arthroplasty — To evaluate Implant survival based on removal or intended removal of any component of the Entrada™ Hip System at five years of follow-up.

SUMMARY:
To evaluate Implant survival based on removal or intended removal of any component of the Entrada™ Hip System at five years of follow-up.

DETAILED DESCRIPTION:
The purpose of this study is to provide clinical evidence for the safety and effectiveness of Ortho Development® Corporation's Entrada™ Hip System (Figure 1). The Entrada™ Hip System was fully introduced to the US market in July, 2018. The Entrada™ Hip System includes the Entrada™ Hip Stem, an FDA approved (510(K) # K171249) femoral stem coupled with either a cobalt chrome or Biolox® Delta Ceramic femoral head. Additionally, the stem and head are coupled with either the Escalade® or Legend® acetabular shell, both of which utilize highly cross-linked polyethylene liners.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo primary total hip arthroplasty using the Entrada™ Hip 2. System due to at least one of the following indications:

* Osteoarthritis
* Inflammatory arthropathy (Rheumatoid Arthritis, Psoriatic Arthritis, etc.) with sufficient bone stock for standard primary THA implants
* Avascular Necrosis with sufficient bone stock for standard primary THA implants
* Post-traumatic Arthritis
* Secondary arthritis due to congenital hip dysplasia 3. Willing and able to provide written informed consent for participation in the study.

  4. Aged 18 - 80 years. 5. Able (in the Investigators opinion) and willing to comply with all study requirements and complete all study visits

Exclusion Criteria:

The potential participant should be excluded from enrollment if any of the following exist:

1. Body mass index ≥ 40
2. History of other orthopaedic surgery within 6 months prior to the index surgery that, in the investigator's opinion, could affect the recovery of the index THA
3. History of pyogenic arthritis in the surgical hip joint
4. Active or suspected infection in or around the surgical hip joint
5. A neurological disorder that, in the investigator's opinion, could affect lower extremity function and recovery from the index THA
6. The potential participant is incarcerated
7. Prior fusion to the index surgical hip joint
8. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

9 . Any other contraindication to THA listed in the Entrada™ Hip Stem Labelling or Instructions for Use.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All orthopaedic patients that are scheduled to undergo primary total hip arthroplasty using the Entrada™ Hip System within 12 weeks will be screened for the following eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-02-28 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Implant Survival | 5 - 10-year follow-up
  Implant survival based on removal or intended removal of any component of Entrada Hip Sys @five years follow-up. Will be measured using the Hip Disability and Osteoarthritis Outcome Score for Joint Reconstruction, the Patient-Reported Outcomes Measurement Information System Global Health Assessment, the UCLA Activity Rating Scale. Effectiveness will be assessed by achieving minimal clinically important difference (MCID) in HOOS JR and UCLA Activity scores. Hung et al. recently reported MCID of HOOS JR to be 19.68 units in an adult recon pop. The MCID for UCLA activity score has been reported to be 0.92 units.minimal detectable change for the PROMIS Global physical and mental health measures will be assessed using one-half of the standard dev between the pre and last post change score. MCID for numeric pain scale will be assessed as a 2 unit change in pain. HOOS, JR score ranges from 1-100 where 0 = total hip disability 100 = perfect hip health.

SECONDARY OUTCOMES:
Implant Survival | 2 - 10 year follow-up
  Implant survival based on removal or intended removal of any component of the Entrada™ Hip System at two and ten years of follow-up. Will be measured using the Hip Disability and Osteoarthritis Outcome Score for Joint Reconstruction (HOOS JR), the PROMIS Global Health Assessment (Physical health, mental health and Numeric pain score), and the UCLA Activity Rating Scale.
Hip Disability and Osteoarthritis Outcome Score for Joint Reconstruction (HOOS JR) | 2 - 10-year follow-up
  The HOOS JR patient reported outcome instrument will be assessed at one, two, five and ten years. The HOOS JR measures function and pain in the involved hip.
PROMIS Global Health Assessment (Physical health, mental health and numeric pain score) | 2 - 10-year follow-up
  The PROMIS Global 10 patient reported outcome instrument will be assessed at one, two, five and ten years. The PROMIS Global 10 measures physical health, mental health and provides an 11 point numeric pain score.
UCLA Activity Rating Scale | 2 - 10-year follow-up
  The UCLA patient reported outcome instrument will be assessed at one, two, five and ten years. The scale is from 1 - 10 with higher values indicating greater physical function.
Patient Satisfaction | 2 - 10-year follow-up
  Patient Satisfaction with their hip replacement will be assessed at one, two, five and ten years. Satisfaction will be measured on a 5 point likert scale from very unsatisfied to very satisfied.
Radiographic Outcomes | 2 - 10-year follow-up
  Radiographic adverse events: Adverse events will be captured on the adverse event case report form. Radiographic adverse events will be evaluated using the zones for radiolucencies as described on the radiographic evaluation case report form. These include the femoral zones described by Gruen et al. Radiolucent lines <2mm will be considered fibrous integration as per the review of Vanrusselt et al. Without evidence of progression these lines will not be considered evidence of aseptic loosening.
Clinical Outcomes | 2 - 10-year follow-up
  Clinical adverse events: Adverse events will be captured on the adverse event case report form.
Patient Satisfaction | 2 - 10-year follow-up
  Satisfaction with the surgical intervention according to the PROMIS Global 10 methods of Rolfson et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health Sciences University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No